CLINICAL TRIAL: NCT05849766
Title: Effect of Dapagliflozin on Cardiac Structure in Patients with Left Ventricular Dysfunction
Brief Title: Effect of Dapagliflozin on Cardiac Structure, Function and Secondary Mitral Regurgitation in Patients with Left Ventricle Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: October 6 University (Other)
Collaborators: National Heart Institute, Egypt (Other Government); University of Florida (Other)
Responsible Party: Principal Investigator, Ahmed Essam, Assistant Lecturer of Clinical Pharmacy, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IHC00044
Record Dates: First submitted 2023-04-27; First posted 2023-05-09 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — dapagliflozin; Ramipril; Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Group 1 received only standard therapy ACE/ ARB, BB, and diuretics
  Interventions: Drug: Ramipril Tritace®, Carvedilol Carvid®,and Spironolactone Aldactone®
- Interventional (Experimental): Group 2 received dapagliflozin 10 mg once daily in addition to standard therapy ACE/ ARB, BB, and diuretics
  Interventions: Drug: Dapagliflozin Farxiga®

INTERVENTIONS:
Drug: Dapagliflozin Farxiga® — Dapagliflozin 10 mg once daily
  Other Names: Forxiga
  Arms: Interventional
Drug: Ramipril Tritace®, Carvedilol Carvid®,and Spironolactone Aldactone® — Ramipril 10 mg once daily, carvedilol 6.25 mg twice daily and spironolactone 25 once daily
  Other Names: Tritace, Carvid, Aldactone
  Arms: Control

SUMMARY:
A significant reduction in the incidence of CV death or hospitalization for HF has been observed in randomized trials investigating the CV benefit of Dapagliflozin. Mechanistic investigations are required to interpret the positive clinical effects of Dapagliflozin on heart structure and valvular regurgitation.

DETAILED DESCRIPTION:
A functional mitral regurgitation (MR) occurs when the mitral valve (MV) becomes tethered due to abnormal LV remodelling in individuals with heart failure (HF) and left ventricular (LV) dilatation.

The primary treatment for HF is medical, and it is based on established guidelines, as LV failure is the most common cause of secondary functional MR. Standard medical therapy for patients with functional MR, including beta blockers, ACE inhibitors, and angiotensin receptor blockers (ARB), does not reduce the morbidity or mortality associated with these conditions.

Similar to the neprilysin inhibitor, which promotes sodium excretion and has vasodilatory effects via relaxing blood vessels, Dapagliflozin reduce cardiac preload and afterload by inducing natriuresis and reducing arterial stiffness. Effects on blood pressure reduction and weight loss may also positively affect left ventricular (LV) remodelling.

Using echocardiography, researchers hope to test the hypothesis that dapagliflozin improves MR in patients with functional MR due to LV dysfunction. This hypothesis is based on studies showing the beneficial effects of Dapagliflozin on LV modelling.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients ≥ 18 years of age
* Dilated LV with a reduced ejection fraction and secondary functional MR
* NYHA functional class II or III
* Moderate to Severe MR which lasted > 6 months under medical treatment with a β-blocker and an ACE inhibitor (or ARB)

Exclusion Criteria:

* Current use or prior use of Dapagliflozin
* Current acute heart failure or prior admission with acute decompensated heart failure in 6 months before entry to study
* NYHA functional class IV
* Chronic renal impairment with GFR < 30 mL/min/1.73m2
* Pregnant or lactating women
* History of allergy to Dapagliflozin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Median / Mean of effective regurgitant orifice area (EROA) of functional mitral regurgitation in patient echocardiographic measures | 6 months
  Change in median / mean of EROA before and after drug administration

SECONDARY OUTCOMES:
Median / Mean of Left ventricle Ejection Fraction (LVEF) of patients in patient echocardiographic measures | 6 months
  Change in median / mean of LVEF before and after drug administration
Median / Mean of Natriuretic peptide concentration (ProBNP) in serum of patients | 6 months
  Change in median / mean of ProBNP before and after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Essam Abou Warda, Principal Investigator — October 6 University
Locations (1):
- Beni-suef University, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No